CLINICAL TRIAL: NCT02990078
Title: Cerebrovascular Reactivity Assessed With Functional Near-infrared Spectroscopy as a Biomarker of Traumatic Microvascular Injury After Moderate-severe Traumatic Brain Injury
Brief Title: Non-invasive Measurement of Cerebrovascular Reactivity After Traumatic Brain Injury
Status: Terminated | Type: Observational
Why Stopped: Sufficient sample size enrolled to demonstrate scientific goals of the study
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Presidential Professor, University of Pennsylvania
Other Study IDs: 825942
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: TBI
Keywords: TBI; CVR; Hypercapnia; fNIRS
MeSH Terms: conditions — Hypercapnia | interventions — Sildenafil Citrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acute TBI: Subjects will be recruited from the neurointensive care unit within 72 hours of their injury. At the time of informed consent, the investigators will perform fNIRS testing with a hypercapnia challenge, fNIRS with hypercapnia challenge 60 minutes after a single oral dose of 50mg sildenafil citrate, outcome qustionaires and symptom checklists (including: Glasgow Outcomes Scale-Extended, Rivermead Post-Concussive Symptom Questionnaire, Brief Symptom Inventory, Alcohol Consumption Questionnaire, Patient Health Questionnaire, and Insomnia Severity Index). This will all be administered again at 14 days, 90 days, 180 days, 1 year, 2 years, 3 years, and 4 years after injury.
  Interventions: Drug: Sildenafil citrate; Device: Functional Near Infared Spectroscopy; Other: Hypercapnia Challenge
- Sub-acute/Chronic TBI: Subjects who suffered a TBI previously and have now entered a subacute or chronic phase of their TBI will be approached by the research team at their clinic visit with a TBI specialist. In those subjects, study timing will be based on the time of their original injury, therefore will start study visits at the next possible time point.
  Interventions: Drug: Sildenafil citrate; Device: Functional Near Infared Spectroscopy; Other: Hypercapnia Challenge
- Healthy Controls: The investigators will also enroll healthy "peer controls". These control subjects will be family members and friends of TBI subjects. These peer controls are likely to have similar environmental and socioeconomic exposures/support which may impact recovery after TBI and may also impact CVR. These control subjects will meet the same inclusion/exclusion criteria as TBI subjects without the requirement for an injury or acute brain imaging. These subjects will be tested in the same way as both TBI groups, but will only have one visit.
  Interventions: Drug: Sildenafil citrate; Device: Functional Near Infared Spectroscopy; Other: Hypercapnia Challenge

INTERVENTIONS:
Drug: Sildenafil citrate — Sildenafil is a potent and specific PDE5 inhibitor, which was initially developed for the treatment of hypertension and angina. Its effectiveness as a treatment for male erectile dysfunction became apparent during Phase I clinical trials, and the focus of drug development shifted to this indication. In patients with cerebrovascular dysfunction, a few preliminary studies have used sildenafil to increase CVR. Participants in the pilot study had CVR tested in response to hypercapnia measured twice, at baseline and then 1 hour after administration of sildenafil citrate, 50 mg by mouth. The investigators have an IND exemption for the uses in this study.
  Other Names: Viagra
Device: Functional Near Infared Spectroscopy — Functional near-infrared spectroscopy (fNIRS) will be used to measure regional cerebral blood flow and cerebrovascular reactivity. are connected to the scalp and surrounding detectors a few cm away detect the light as it scatters through the underlying tissues. The technique is able to detect changes in the absorption spectrum of the tissue corresponding to the concentrations of oxyhemoglobin (HbO2) and deoxyhemoglobin (HbR), and indicate local perfusion changes.
  Other Names: fNIRS
Other: Hypercapnia Challenge — The study device is a Douglas Bag that traditionally is designed to measure respiratory exchange. It consists of large bag attached to a mouthpiece utilized to hold either expired air from the subject or filled with different concentrations of air to be aspired. For the purposes of this study, the Douglas Bag will be utilized to induce hypercapnia in the subject. The bag is equipped with a switch that allows rapid shifting from room air to 5% CO2 each minute over 7 minutes.

SUMMARY:
The investigators will longitudinally measure cerebrovascular reactivity (CVR) by functional near-infrared spectroscopy (fNIRS) in acute (≤3 days from injury), subacute, and chronic phases after TBI as a biomarker of TCVI as compared to healthy controls. CVR will be measured by fNIRS response to hypercapnia. The investigators hypothesize that CVR will be decreased after TBI and that these decreases will correlate with clinical outcomes. Furthermore, the investigators predict that administration of a vasodilatory medication (sildenafil) will augment CVR after TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged ≥18
2. CT evidence of TBI-linked abnormality

   * Traumatic subarachnoid hemorrhage
   * Intracerebral hemorrhage/contusion
   * Subdural/epidural hematoma
3. Ability to undergo fNIRS testing with hypercapnia challenge
4. Subject able to provide informed consent
5. Attending of record agrees to include subject in study

Exclusion Criteria:

1. Unstable respiratory or hemodynamic status
2. Evidence of penetrating brain injury
3. TBI requiring craniotomy or craniectomy
4. Evidence or risk of ICP crisis
5. History of disabling pre-existing neurologic disorder (e.g. dementia, uncontrolled epilepsy, multiple sclerosis, strokes, brain tumors, prior severe TBI, or other disorder that confounds interpretation of NIRS testing or neuropsychological results)
6. History of pre-existing disabling mental illness (e.g. major depression or schizophrenia)
7. Exclusion criteria for sildenafil administration:

   * History of melanoma
   * current use of organic nitrate vasodilators
   * current use of ritonavir (HIV-protease inhibitor)
   * current use of erythromycin, ketoconazole, or itraconazole; current use of cimetidine
   * current use of alpha-blockers such as doxazosin (Cardura), tamsulosin (Flomax), and terazosin (Hytrin) prazosin (Minipres)
   * resting hypotension (systolic BP <90)
   * severe renal insufficiency
   * hepatic cirrhosis
   * acute ischemic stroke within past 2 months
   * acute myocardial infarction within past 2 months
   * unstable angina pectoris
   * acute or chronic heart failure
   * retinitis pigmentosa
   * pregnant or breastfeeding female
   * known hypersensitivity or allergy to sildenafil
8. Unstable cardiac status that constitutes a contraindication to sexual activity
9. Inability to read and communicate in English (necessary to obtain reliable neuropsychometric data)
10. Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female, aged 18 or older, presenting with a diagnosis of traumatic brain injury (TBI) and healthy peer control volunteers .
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in CVR prior to sildenafil administration | < 72hrs, 14 days, 90 days, 180 days, 1 year, 2 years, 3 years, 4 years

SECONDARY OUTCOMES:
Change CVR after sildenafil administration | <72 hours, 14 days, 90 days, 180 days, 1 year, 2 years, 3 years, 4 years
Relationship of CVR with symptom reports, as measured by the Neurobehavioral Symptom Inventory (NBSI). | < 72hrs, 14 days, 90 days, 180 days, 1 year, 2 years, 3 years, 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Diaz-Arrastia, MD, PhD, Principal Investigator — University of Pennsylvania Perelman School of Medicine, Department of Neurology
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No